CLINICAL TRIAL: NCT03859609
Title: Failure Prediction of Adult Spinal Deformity Surgery Comparing GAP-score With Schwab-score
Brief Title: Comparison of GAP-score With Schwab-score
Status: Completed | Type: Observational
Sponsor: Mohammad ARAB MOTLAGH (Other)
Responsible Party: Sponsor-Investigator, Mohammad ARAB MOTLAGH, MD, PhD, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Other Study IDs: Adult Spinal Deformity Surgery
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Spinal Fusion; Adjacent Segment Degeneration
Keywords: GAP-score; Schwab score; Proximal Junctional Failure; Spinal Fusion
MeSH Terms: interventions — Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Spinal Fusion — Spinal alignment was evaluated according to two different score-systems

SUMMARY:
The predictive value of two different score-systems with regard to failure rate following long extent spinal fusion is subject of evaluation.

DETAILED DESCRIPTION:
The multilevel spinal fusion is associated with high rate of failure. This results from insufficient adaptation of the fused spine to the proper individual spinal alignment. In the recent years, comprehensive understanding of spinal alignment and definition of several parameters contributed to develop score systems to evaluate the alignment of the multilevel spinal fusion and to predict failure. In the following study the results of multilevel spinal fusion were evaluated retrospectively according to two scoring systems: GAP-score und Schwab-score. The predictive value of each score system is analyzed by the correlation of the failure rate with its corresponding score value.

ELIGIBILITY:
Inclusion Criteria:

* 3 and more fusion levels

Exclusion Criteria:

* Neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had fusion operation with dorsal instrumentation on at least 3 spinal levels
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Radiological Evaluation | 2 months
  Pelvic tilt in degree, Pelvic incidence in degree, Sacral slope in degree, Lumbar lordosis in degree, L5-S1 lordosis in degree, Thoracic kyphosis in degree, Sagittal vertical axis in degree, Thoracolumbar kyphosis in degree, Global tilt in degree, Cobb angle in degree

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Arab Motlagh, MD, PhD, Principal Investigator — Goethe University
Locations (1):
- Department of Orthopaedic Surgery, University Hospital Frankfurt, Frankfurt, Germany